CLINICAL TRIAL: NCT02908334
Title: Sertraline in Addition to Standard of Care Treatment for Coccidioidomycosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: failure to enroll
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UCSF-Fresno-01
Record Dates: First submitted 2016-09-14; First posted 2016-09-20 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Coccidioidomycosis
MeSH Terms: conditions — Coccidioidomycosis | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): standard of care treatment for disseminated or meningeal coccidioidomycosis
- Standard of Care + Sertraline (Experimental): Standard of care treatment with the addition of sertraline for the treatment of disseminated or meningeal coccidioidomycosis
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline — 400 mg/day sertraline
  Arms: Standard of Care + Sertraline

SUMMARY:
In this study patients will be randomized 1:2 to receive either standard of care treatment or standard of care + Sertraline 200mg/day for 2 weeks, then 400 mg/day for 50 weeks for treatment of disseminated and meningeal coccidioidomycosis.

DETAILED DESCRIPTION:
Sertraline has been demonstrated to have in-vitro activity against coccidioides, and in-vivo activity against cryptococcal meningitis in clinical trials. Disseminated and meningeal coccidiodes infections require lifelong treatment, have poor outcomes, and new treatment options are needed. In this study the investigators will determine safety and tolerability of adjunctive sertraline (grade 4-5 adverse reactions) compared to standard coccidioidomycosis therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Severe coccidioidomycosis infection, manifest as by one of:

  * Coccidioidal meningitis;
  * Severe pulmonary infection requiring intensive care unit level of care;
  * Disseminated infection (in clinical opinion of the investigator); or
  * Clinical progression after >2 months of high dose fluconazole.
* Laboratory confirmation of Coccidioides infection by culture, histopathology, coccidioides polymerase chain reaction, positive complement fixation titer, or Coccidioides antigen

Exclusion Criteria:

* Age < 18 years
* Cannot or unlikely to attend regular clinic visits
* Presence of jaundice or known liver cirrhosis
* Pregnancy

  * If there is a concern of pregnancy, a negative urine (or serum) pregnancy test before study entry is required.
  * Women of childbearing potential will have pregnancy test at enrollment and will be recommended to use contraception and referred to family planning services as necessary. (Refer to informed consent document.)
* Currently breastfeeding
* Active drug use (amphetamine or cocaine) or requirement for concomitant medications that raise the risk of serotonin syndrome
* Prolonged corrected QT interval or Left Bundle Branch Block on baseline electrocardiogram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Adverse Reactions | 2 years
  grade 4-5 adverse reactions

SECONDARY OUTCOMES:
Mycoses Study Group Score | 2 years
  scoring of clinical outcomes
Depression Screening | 2 years
  Patient Health Questionnaire 9
Functional Assessment | 2 years
  Karnofsky

CONTACTS AND LOCATIONS:
Overall Officials: Simon Paul, MD, Principal Investigator — UCSF - Fresno

IPD SHARING:
Plan to Share IPD: No